CLINICAL TRIAL: NCT06932666
Title: Why Calories Are Not the Same - a Gut Explanation
Brief Title: Why Calories Are Not the Same - a Gut Explanation?
Acronym: GutEnergy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Henrik Munch Roager, Associate Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M408
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-04

CONDITIONS: Diet, Healthy; Breath Analysis
Keywords: Fecal energy; Metabolizable energy; Breath methane; Gut microbiome; Metabolomics; Dietary fiber; Resistant starch; Food particle size

STUDY DESIGN:
Intervention Model Description: Overall, there are two parallel arms - high- (HMP) and low- (LMP) methane producers, to which the participants are allocated in a ratio 1:1 after a 4-day screening period, where individual levels of methane in exhaled breath are measured multiple times.
  In both arms, participants undergo two 3-days dietary interventions in a crossover design and separated by a +10-day washout period. Participants are randomized to receiving diet A first or diet B first. These two diets are isocaloric and equal in macronutrient composition, but differ on dietary fiber, resistant starch and food particle size.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-methane producers (Experimental): Individuals exhaling high levels of methane (median exhaled methane >= 5 ppm), as measured 3-times daily during the screening period.
  Interventions: Other: Diet A group; Other: Diet B group
- Low-methane producers (Experimental): Individuals exhaling low levels of methane (median exhaled methane < 5 ppm), as measured 3-times daily during the screening period.
  Interventions: Other: Diet A group; Other: Diet B group

INTERVENTIONS:
Other: Diet A group — Diet high in fiber (> 40g/10MJ), high in resistant starch (> 10g/10MJ), and containing large food particles. Diet is provided for 3 full days, consists of three meals per day (breakfast, lunch, and dinner) and in-between meals, and covers 100% of the participants' energy requirements.
Other: Diet B group — Diet low in fiber (< 10g/10MJ), low in resistant starch (< 3g/10MJ) and containing small food particles. Diet is provided for 3 full days, consists of three meals per day (breakfast, lunch, and dinner) and in-between meals, and covers 100% of the participants' energy requirements.

SUMMARY:
The aim of this study is to understand how the gut microbiome influences how much dietary energy humans excrete via feces. This study is based on the hypothesis that levels of methane in exhaled breath represent two different gut microbiome community structures, and therefore influence fecal energy excretion differently. Moreover, this study is assessed in the context of two different diets, both isocaloric and equal in macronutrient composition, but differing in contents of fiber, resistant starch, and large particles; which are hypothesized to impact the gut microbiome differently.

DETAILED DESCRIPTION:
The trial is a cross-over trial including two controlled isocaloric dietary interventions of three days duration. The two diets are isocaloric but with different contents of fiber, resistant starch, and food particle sizes. Each intervention is separated by a wash-out period of at least 10 days where participants adhere to their habitual diet. The trial includes a total of five visits (one screening visit and four regular visits).

Before the trial, participants undergo a screening period of 4 days. During the 4-day screening period, participants measure the levels of methane in their exhaled breath. Based on median breath methane levels, participants are allocated to one of the two arms: (HMP: high methane producers; LMP: low methane producers). Enrollment in the intervention trial will be conducted so there are similar numbers of participants in both arms.

At the beginning and at the end of each 3-day intervention period, participants consume a blue muffin, containing a royal blue dye that changes the stool color. The appearance of the color in stool following the first muffin will mark the beginning of the stool collection period, which will continue until the stool color change is no longer noticeable following consumption of the second muffin. Therefore, the duration of the stool collection period, which is estimated to be on average 3 days, will ultimately depend on the participants' passage time of food (i.e., intestinal transit time).

During the screening period, participants are asked to:

* measure their methane and hydrogen levels in exhaled breath using a portable device
* report defecation patterns (including stool frequency and Bristol Stool Scale)

Before each intervention period, participants are asked to:

* collect a fecal and urine sample
* register three days of habitual diet

At the visits before each intervention period, the following samples are collected:

* a blood sample
* methane and hydrogen measurements in exhaled breath
* anthropometrics
* data on physical activity

During the intervention periods, participants are asked to:

* exclusively eat all the foods provided
* collect all their stool samples, as specified above
* collect three morning urine samples (one daily for the following three days)
* measure their methane and hydrogen levels in their exhaled breath using a portable device
* report their defecation patterns and gastrointestinal symptoms

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* BMI:18.5-29.9 kg/m2
* Self-reported regular defecations defined as at least every second day
* Willing to collect urine and stool samples at home and able to temporarily store them in their own freezer in a provided container
* Willing to exclusively eat the food provided
* Owning a smartphone (iOS 11.0 and onwards, or Android 5.0 and onwards) with access to the internet
* Speak and understand Danish or English

Exclusion Criteria:

* Current pregnancy or lactation
* Following a specific dietary program or diet (e.g., vegetarian, vegan, gluten-free) or unable to consume the food provided
* Diagnosis of small intestinal bacterial overgrowth (SIBO), inflammatory bowel diseases (IBD), gastrointestinal obstruction, or ischemic colitis
* Diagnosed chronic constipation
* Regular use of diarrhea inhibitors or laxatives
* Any chronic disease that can affect the outcomes of the study
* Use of medications potentially altering gastric pH (proton pump inhibitors, histamine receptor antagonists, antacids)
* Use of medications potentially altering the gastro-intestinal motility (prokinetics, antiemetic agents, anticholinergic agents, narcotic analgesics, nonsteroidal anti-inflammatory drugs, peroral glucocorticoids, and GLP-1 related medications such as semaglutide and liraglutide)
* Use of antibiotics, or any medication that can affect any outcomes of the study, within the previous three months
* Concurrent participation in another trial
* Any condition that makes the project responsible and/or the clinical responsible doubt the feasibility of the volunteer's participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total fecal energy excretion (between high- and low-methane producers) | During each stool collection period (following each 3-day intervention period)
  Differences in total fecal energy excretion, determined as total kilocalories excreted via feces, between low and high methane producers following intake of the two controlled, isocaloric diets.

SECONDARY OUTCOMES:
Total fecal energy excretion (between diet A and diet B) | During each stool collection period (following each 3-day intervention period)
  Differences in total fecal energy excretion, determined as total kilocalories excreted via feces, between the two isocaloric diets (that differ in fiber, resistant starch, and particle size).
Fecal energy density | During each 3-day intervention period and its following stool collection period
  Differences in fecal energy density, determined as fecal energy (kcal) relative to fecal weight, between high- and low-methane producers.
Total fecal weight excreted | During each 3-day intervention period and its following stool collection period
  Differences in total fecal weight excreted, determined as dry weight (grams), between high- and low-methane producers.
Breath hydrogen and methane levels | During each 3-day intervention period and its following stool collection period
  Differences in breath methane and hydrogen concentration in exhaled breath, measured in parts per million (PPM), between high- and low-methane producers.
Whole-gut transit time | During each 3-day intervention period and its following stool collection period
  Differences in whole-gut transit time, determined by the passage time of muffins with blue dye, between high- and low-methane producers.
Stool consistency | During each 3-day intervention period and its following stool collection period
  Differences in stool consistency, determined by Bristol Stool Scale, between high- and low-methane producers.
Stool frequency | During each 3-day intervention period and its following stool collection period
  Differences in stool frequency, determined by defecation records registered by the participants, between high- and low-methane producers.
Stool moisture | During each 3-day intervention period and its following stool collection period
  Differences in stool moisture, determined as fecal water content relative to fecal weight, between high- and low-methane producers.
Fecal pH | During each 3-day intervention period and its following stool collection period
  Differences in fecal pH between high- and low-methane producers.
Fecal microbial load | During each 3-day intervention period and its following stool collection period
  Differences in fecal microbial load, determined as total microbial DNA reads in feces, between high- and low-methane producers.
Fecal host DNA concentration | During each 3-day intervention period and its following stool collection period
  Differences in fecal host DNA concentration, determined as total human DNA reads in feces, between high- and low-methane producers.
Fecal short-chain fatty acids | During each 3-day intervention period and its following stool collection period
  Differences in fecal short-chain fatty acid concentrations between high- and low-methane producers.
Gut microbiome composition (16S) | During each 3-day intervention period and its following stool collection period
  Differences in gut microbiome composition, determined by 16S amplicon sequencing of fecal DNA, between high- and low-methane producers.
Gut microbiome composition and functions (shotgun sequencing) | During each 3-day intervention period and its following stool collection period
  Differences in gut microbiome taxonomic composition and functions, determined by shotgun sequencing of fecal DNA, between high- and low-methane producers.

OTHER OUTCOMES:
Gut microbiome-derived metabolites (fecal samples) | During each 3-day intervention period and its following stool collection period
  Differences in gut microbiome-derived metabolites, such as short-chain fatty acids, bile acids, amino acid-derived metabolites, and other metabolites derived from microbial proteolytic and saccharolytic fermentation measured from fecal samples, between high- and low-methane producers.
Gut microbiome-derived metabolites (urine samples) | Before and during each 3-day intervention period
  Differences in gut microbiome-derived metabolites, such as short-chain fatty acids, bile acids, amino acid-derived metabolites, and other metabolites derived from microbial proteolytic and saccharolytic fermentation measured from urine samples, between high- and low-methane producers.
Gut microbiome-derived metabolites (blood samples) | Right before each 3-day intervention period
  Differences in gut microbiome-derived metabolites, such as short-chain fatty acids, bile acids, amino acid-derived metabolites, and other metabolites derived from microbial proteolytic and saccharolytic fermentation measured from blood samples, between high- and low-methane producers.
Fecal metabolome (untargeted metabolomics) | During each 3-day intervention period and its following stool collection period
  Differences in the fecal metabolome, measured by LC-MS/MS untargeted metabolomics, between high- and low-methane producers.
Urine metabolome (untargeted metabolomics) | Before and during each 3-day intervention period
  Differences in the urine metabolome, measured by LC-MS/MS untargeted metabolomics, between high- and low-methane producers.
Blood metabolome (untargeted metabolomics) | Right before each 3-day intervention period
  Differences in the blood metabolome, measured by LC-MS/MS untargeted metabolomics, between high- and low-methane producers.
Gastrointestinal symptoms | During each 3-day intervention period
  Differences in the gastrointestinal symptoms during the 3-day intervention period, measured using a visual analog scale, between high- and low-methane producers.
Habitual diet records | Right before each 3-day intervention period
  Differences in habitual diet records registered by participants, between high- and low-methane producers.
Habitual physical activity records | Baseline (before the first 3-day intervention period)
  Differences in habitual physical activity records registered by participants, between high- and low-methane producers.
Body weight | Right before each 3-day intervention period
  Differences in body weight before intervention, between high- and low-methane producers.
Body fat composition | Baseline (before the first 3-day intervention period)
  Differences in body fat composition, measured through Dual-Energy X-ray Absorptiometry (DXA scan), between high- and low-methane producers.
Muscle composition | Baseline (before the first 3-day intervention period)
  Differences in muscle composition, measured through Dual-Energy X-ray Absorptiometry (DXA scan), between high- and low-methane producers.
Bone composition | Baseline (before the first 3-day intervention period)
  Differences in bone composition, measured through Dual-Energy X-ray Absorptiometry (DXA scan), between high- and low-methane producers.
Biomarkers of food intake (fecal samples) | During each 3-day intervention period and its following stool collection period
  Differences in biomarkers of food intake, measured by untargeted metabolomics and food DNA in fecal samples, between high- and low-methane producers.
Biomarkers of food intake (urine samples) | Before and during each 3-day intervention period
  Differences in biomarkers of food intake, measured by untargeted metabolomics in urine samples, between high- and low-methane producers.
Biomarkers of food intake (blood samples) | Right before each 3-day intervention period
  Differences in biomarkers of food intake, measured by untargeted metabolomics in blood samples, between high- and low-methane producers.
Fecal particle size | During each 3-day intervention period and its following stool collection period
  Differences in fecal particle size between high- and low-methane producers.
Fecal carbon-to-nitrogen ratio | During each 3-day intervention period and its following stool collection period
  Differences in fecal carbon-to-nitrogen ratio between high- and low-methane producers.
Fecal redox potential | During each 3-day intervention period and its following stool collection period
  Differences in fecal redox potential, measured in millivolts (mV), between high- and low-methane producers.
Fecal biomarkers of inflammation: calprotectin | During each 3-day intervention period and its following stool collection period
  Differences in fecal biomarkers of inflammation, determined by fecal calprotectin, between high- and low-methane producers.
Fecal biomarkers of intestinal permeability: zonulin | During each 3-day intervention period and its following stool collection period
  Differences in fecal biomarkers of intestinal permeability, determined by fecal zonulin, between high- and low-methane producers.
Blood markers of glucose metabolism | Right before each 3-day intervention period
  Differences in blood markers of glucose metabolism, such as glucose, insulin and HbA1C, between high- and low-methane producers.
Blood markers of lipid metabolism | Right before each 3-day intervention period
  Differences in blood markers of lipid metabolism, such as total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglycerides, between high- and low-methane producers.
Blood markers of inflammation | Right before each 3-day intervention period
  Differences in blood markers of inflammation, such as CRP, IL-6, TNF-α, and other cytokines, between high- and low-methane producers.
Blood markers of appetite | Right before each 3-day intervention period
  Differences in blood markers of appetite, such as glucagon, GLP-1, GLP-2, PYY, leptin, ghrelin, GIP, and CCK, between high- and low-methane producers.
Blood markers of intestinal permeability: LBP | Right before each 3-day intervention period
  Differences in blood markers of intestinal permeability, such as lipopolysaccharide-binding protein (LBP), between high- and low-methane producers.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Department of Nutrition, Exercise and Sports, Frederiksberg, Capital Region, Denmark